CLINICAL TRIAL: NCT02365441
Title: A Randomised Phase II Trial of Imatinib Alternating With Regorafenib Compared to Imatinib Alone for the First Line Treatment of Advanced Gastrointestinal Stromal Tumour (GIST)
Brief Title: A Randomised Trial of Imatinib Alternating With Regorafenib Compared to Imatinib Alone for the First Line Treatment of Advanced Gastrointestinal Stromal Tumour (GIST)
Acronym: ALT GIST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Scandinavian Sarcoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG1013GST; ACTRN12614000950662 (Other: ANZCTR)
Record Dates: First submitted 2014-11-04; First posted 2015-02-19 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Stromal Tumour
Keywords: GIST; Advanced
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): imatinib 400mg orally daily continuously
  Interventions: Drug: imatinib
- Arm B (Experimental): alternating 28-day periods of imatinib 400mg orally daily for 21 to 25 days followed by a washout (drug free) period of 3 to 7 days, then regorafenib 160mg orally daily for 3 weeks followed by a 7 day washout (drug free) period.
  Interventions: Drug: Regorafenib; Drug: imatinib

INTERVENTIONS:
Drug: Regorafenib
  Arms: Arm B
Drug: imatinib
  Other Names: Glevec

SUMMARY:
An open label randomised trial for adults with histologically confirmed measurable metastatic GIST who have received no other treatment for metastatic disease. The study aims to determine if an alternating regimen of imatinib and regorafenib has sufficient activity and safety in comparison to imatinib alone to warrant further evaluation as a first line treatment for metastatic GIST.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS Background Despite highly active current treatment for metastatic gastrointestinal stromal tumour (GIST) with the use of imatinib, most people will ultimately relapse and die of multifocal metastatic disease. Using an alternating regimen of imatinib and regorafenib with brief drug free intervals may allow tumour stem cells to re-enter the cell cycle and become susceptible once more to drug therapy. Regorafenib, a multi-targeted tyrosine kinase inhibitor (TKI) with activity against angiogenic, stromal and oncogenic receptor tyrosine kinases, has demonstrated activity in the treatment of GIST and is FDA approved for third line therapy of advanced GIST.

General aim To determine if an alternating regimen of imatinib and regorafenib has sufficient activity and safety to warrant further evaluation as a first line treatment for metastatic GIST.

Design Prospective, randomised, open label phase II trial, stratified by participating site, previous adjuvant therapy (prior vs none), and previous imatinib for metastatic disease for less than 21 days.

Population The target population is adults with histologically confirmed, measurable metastatic GIST, who have received no prior treatment for metastatic disease. Patients who are currently taking, and have had up to 21 days of uninterrupted treatment with 400mg daily of imatinib are eligible to participate in this study.

Study treatments

Patients will be randomised to receive either:

Arm A - imatinib 400mg orally daily continuously (control arm); or Arm B - alternating 28-day periods of imatinib 400mg orally daily for 21 to 25 days followed by a washout (drug free) period of 3 to 7 days, then regorafenib 160mg orally daily for 3 weeks followed by a 7 day washout (drug free) period.

Treatment will continue until disease progression or prohibitive adverse events as detailed in the protocol.

Statistical considerations In order to demonstrate a relative increase in progression free survival at 24 months from the date of randomisation from an expected 78% to 88%, with 80% power and 95% confidence based on A'Hern's adjustment to Fleming's design, approximately 110 evaluable participants will be required in each arm. Thus, it is proposed to enrol 240 participants into the trial, allowing for approximately a 10% drop-out rate. Currently 80% of participants are expected to achieve a clinical benefit at 24 months (CBR - rate of complete or partial response, or stable disease). A secondary outcome would be to determine whether a minimum 25% relative increase of the CBR (from 80% to 85%) in the experimental cohort can be attained. The study will be open to recruitment for 36 months while follow-up will continue until the last enrolled participant has been followed for a minimum of 24 months timed from the date of commencement of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 yrs) with histologically confirmed GIST. In CD-117-negative cases DOG-1 must be positive or a KIT/PDGFRA mutation must be present.
* Unresectable, metastatic disease.
* No prior TKI for metastatic disease, with the exception of those patients who have had up to 21 days of uninterrupted treatment on 400mg daily of imatinib.
* Imatinib therapy given as an adjuvant treatment and completed at least 3 months prior to entry into this trial is permitted. Patients who have progression of GIST while on adjuvant therapy are not eligible for this trial.
* ECOG performance status 0-2
* Measurable disease by RECIST version 1.1. (Note: Participants with only peritoneal disease will be eligible only if they have lesions measurable in two dimensions and have at least 1 lesion which is ≥ 2 cm in size).
* Adequate bone marrow function (Haemoglobin ≥ 9.0g/dL, platelet count ≥ 100 x 109/L, and absolute neutrophil count ≥ 1.5 x 109/L).
* Adequate liver function (Serum total bilirubin ≤1.5 x ULN, INR ≤ 1.5, and ALT, AST, ALP ≤2.5 x ULN (≤ 5 x ULN for participants with liver metastases). Lipase level must be ≤ 1.5 x ULN.
* Adequate renal function (Creatinine clearance > 50ml/min) based on either the Cockcroft Gault formula, 24 hour urine or Glomerular Filtration Rate (GFR scan); and serum creatinine ≤ 1.5 x ULN.
* Tumour tissue available for central review.
* Willing and able to comply with all study requirements, including treatment timing and/or nature of required assessments.
* Study treatment both planned and able to start within 14 days of randomisation.
* Signed, written informed consent.

Exclusion Criteria:

* Concurrent GI illness which may prevent absorption of imatinib or regorafenib - please note that prior gastrectomy or bowel resection does not exclude patients from this study.
* Use of other investigational drugs within 4 weeks prior to enrolment.
* Known sensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
* Participants receiving therapeutic doses of warfarin.
* Presence of brain metastases.
* The presence of PDGFR D842V mutation or other mutation known to cause imatinib resistance.
* Inability to swallow tablets.
* Arterial thrombotic or ischaemic events, such as cerebrovascular accident or pulmonary embolism within 6 months prior to randomisation; or major venous thrombotic events requiring use of an anticoagulant such as warfarin within 6 months prior to randomisation.
* Poorly controlled hypertension (systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomisation, or non healing wound, ulcer or fracture.
* Congestive cardiac failure (NYHA ≥ grade 2), unstable angina or new onset angina within the previous 3 months, or AMI within the previous 6 months. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Haemorrhage or bleeding event ≥ Grade 3 according to CTCAE v4.0 within 4 weeks prior to randomisation.
* Ongoing infection of > Grade 2 according to CTCAE v4.0.
* Active hepatitis B or C or HIV, or chronic hepatitis B or C requiring treatment with antiviral therapy. Testing for these is not mandatory unless clinically indicated.
* Interstitial lung disease with ongoing signs and symptoms.
* Persistent proteinuria of ≥ Grade 3 (>3.5g/24 hours) according to CTCAE v4.0
* Other significant medical or psychiatric condition judged by the investigator to interfere with protocol requirements.
* Use of biological response modifiers such as granulocyte colony stimulating factor (G-CSF), within 3 weeks prior to randomisation.
* Patients taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinovir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg carbamazepine, phenobarbitol, phenytoin, rifampicin, St John's wort).
* History of another malignancy within 5 years prior to registration. Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 5 years after definitive primary treatment.
* Pregnancy, lactation, or inadequate contraception. Women must be post menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Women of childbearing potential and men must agree to use adequate contraception before entering the trial until at least 8 weeks after the last study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective tumour response (complete or partial response) as determined by RECIST v1.1 | At or before 9 months from the time from either (i) randomization (if patients have not yet commenced treatment) or (ii) commencement of therapy (if patients are randomized during the first cycle of imatinib)
  The objective tumour response rate (OTRR) will be calculated by summing the number of participants assessed as having a complete or partial response within the first 9 months from the time from either (i) randomization (if patients have not yet commenced treatment) or (ii) commencement of therapy (if patients are randomized during the first cycle of imatinib), and dividing this by the total number of participants evaluable for response. For patients who undergo surgery, the best response is determined in the time period that precedes the date of surgery. The responses are confirmed at the time of the next scheduled imaging, usually done 8 weeks after the first detection of response, provided that imaging of the target lesions is not indicated sooner than this for other reasons. Both the numbers and the proportions of confirmed and unconfirmed responses will be reported. The minimum duration of SD is defined as 8 weeks.

SECONDARY OUTCOMES:
Progression free survival at 24 months (disease progression or death) | 24 Months
  PFS at 24 months as calculated from the time from either (i) randomization if patients have not yet commenced treatment) or (ii) commencement of therapy (if patients are randomized during the first cycle of imatinib) to the date of progression as determined by RECIST v1.1
Clinical benefit rate at 24 weeks | 24 weeks
  Clinical benefit rate (SD + PR + CR) following 2 cycles of treatment
Time to treatment failure | 5 years
  Time to treatment failure is defined as the time from either (i) randomization (if patients have not yet commenced treatment) or (ii) commencement of therapy (if patients are randomized during the first cycle of imatinib) to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.
Adverse Events | 5 years
  Safety/toxicity/tolerability
Overall survival | 5 years
  Overall survival is defined as the interval from either (i) randomization (if patients have not yet commenced treatment) or (ii) commencement of therapy (if patients are randomized during the first cycle of imatinib) to date of death from any cause, or the date of last known follow-up alive.

OTHER OUTCOMES:
Macroscopically complete removal of all residual disease by surgery | 5 years
  This is defined as the rate of patients who proceed to surgery with the aim of resecting all remaining macroscopic disease.
Change in PET imaging during washout period of regorafenib and imatinib in those taking part in the PET substudy | 3 years
  to explore the relationship between change in PET imaging during washout period of regorafenib and imatinib (in subset of participants at selected centres)
Imatinib plasma levels 4 and 12 weeks after commencement of treatment in both arms. Arm B: Imatinib plasma levels at 3 and 11 weeks after commencement of treatment and regorafenib plasma levels 7 and 15 weeks after commencement of treatment. | 3 years
  To explore the relationship between study endpoints and Imatinib plasma levels at 4 and 12 weeks after commencement of treatment in both arms. Arm B: Imatinib plasma levels at 3 and 11 weeks after commencement of treatment and regorafenib plasma levels 7 and 15 weeks after commencement of treatment.
Change in circulating serum/plasma growth factor and cytokine levels over time(multiplex assay), Frequency of KIT/PDGFRA mutations in circulating blood DNA and DNA load as prognostic and/or predictive markers | 3 years
  To explore the relationship between study endpoints and circulating other biomarkers as prognostic and/or predictive markers.
Tumour tissue biomarkers including, but not limited to, proteins relating to EGFR and PDGFR signalling and angiogenesis. | 3 years
Macroscopically complete removal of all residual disease by surgery | 3 years
  Rate of patients having macroscopically complete removal of all residual disease by surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, Professor, Study Chair — SSG; Desmond Yip, A/Professor, Study Chair — AGITG
Locations (25):
- Australia (10):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Calvary Mater Newcastle Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Ashford Cancer Centre Research, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner, Perth, Western Australia
- Helsinki University Hospital, Helsinki, Finland
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Léon
  - Institut Gustave Roussy, Paris
- Netherlands Cancer Institute -Antoni Van Leeuwenhoek, Amsterdam, Netherlands
- Norway (2):
  - Haukeland University Hospital, Bergen
  - The Norwegian Radium Hospital, Oslo
- National Cancer Centre Singapore, Singapore, Singapore
- National Cancer Institute, Bratislava, NSW, Slovakia
- ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona, Spain
- Lund University Hospital, Lund, Sweden
- United Kingdom (3):
  - University Hospital Birmingham - Queen Elizabeth Hospital, Birmingham
  - Royal Marsden Hospital, London
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham

REFERENCES:
- [Derived] Yip D, Zalcberg J, Blay JY, Eriksson M, Espinoza D, Price T, Marreaud S, Italiano A, Steeghs N, Boye K, Underhill C, Gebski V, Simes J, Gelderblom H, Joensuu H. Imatinib alternating with regorafenib compared to imatinib alone for the first-line treatment of advanced gastrointestinal stromal tumor: The AGITG ALT-GIST intergroup randomized phase II trial. Br J Cancer. 2025 Jun;132(10):897-904. doi: 10.1038/s41416-025-02983-w. Epub 2025 Mar 25. PMID 40133509